CLINICAL TRIAL: NCT05200507
Title: Physiological Effects on Lung Aeration of High Frequency Percussive Ventilation in Hypersecretive Tracheostomized Patients: a Physiological Observational Study
Brief Title: High Frequency Percussive Ventilation in Hypersecretive Tracheostomized Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Prof, University Magna Graecia
Other Study IDs: Percussionaire-tracheo
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Acute Respiratory Failure; Pneumonia
Keywords: Secretions; tracheostomized critically ill patients
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High frequency precussive ventilation: After positioning a silicon belt for Electrical Impedance Tomography (EIT) and a baseline record, patients will receive the treatment of High Frequency Percussive Ventilation. Further recordings will be acquired soon after the end of the treatment, 1 and 3 hours later.
  Interventions: Device: High Frequency Percussive Ventilation

INTERVENTIONS:
Device: High Frequency Percussive Ventilation — High Frequency Percussive Ventilation will be applied for 10 minutes at an oscillation frequency of 10 Hz, superimposed to the ventilatory assistance

SUMMARY:
The incidence of pulmonary complications such as pulmonary atelectasis, pneumonia (including ventilator-associated pneumonia), and acute respiratory failure is high in critical care patients. The incidence of ventilator-associated pneumonia can be as high as 27% amongst mechanically ventilated patients. Studies have shown that 16% of critically ill patients have been reported to develop acute respiratory failure, which is associated with prolonged intensive care unit stay, resulting in significantly higher mortality than non-respiratory failure patients. Increased morbidity and mortality contribute to the burden on the health care system and lead to poor health-related outcomes. Multimodal physiotherapy plays a role in the management of these critically ill patients. High frequency percussive ventilation (HFPV) is used in patients with underlying pulmonary atelectasis, excessive airway secretions, and respiratory failure. HFPV is a non-continuous form of high-frequency ventilation delivered by a pneumatic device that provides small bursts of sub-physiological tidal breaths at a frequency of 60-600 cycles/minute superimposed on a patient's breathing cycle. The high-frequency breaths create shear forces causing dislodgement of the airway secretions. Furthermore, the HFPV breath cycle has an asymmetrical flow pattern characterized by larger expiratory flow rates, which may propel the airway secretions towards the central airway. In addition, the applied positive pressure recruits the lung units, resulting in a more homogeneous distribution of ventilation and improved gas exchange. In acute care and critical care settings, HFPV intervention is used in a range of patients, from spontaneously breathing patients to those receiving invasive mechanical ventilation where HFPV breaths can be superimposed on a patient's breathing cycle or superimposed on breaths delivered by a mechanical ventilator. The most common indications for HFPV use are reported as removal of excessive bronchial secretions, improving gas exchange, and recruitment of atelectatic lung segments. This study aims to assess the lung physiological response to HFPV in terms of aeration and ventilation distribution.

ELIGIBILITY:
Inclusion Criteria:

* more than 48 hours of invasive mechanical ventilation
* presence of tracheostomy
* need for two or more broncoaspirations per hour in the previous 8 hours

Exclusion Criteria:

* life threatening cardiac arrythmia
* pneumothorax
* acute spinal injury
* chest trauma
* brain injury in the previous 15 days
* hemodynamic instability
* chest or abdominal surgery in the previous 7 days
* pregnancy
* enrollment in other study protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All tracheostomized patients requiring invasive mechanical ventilation for more than 48 hours and with an hypersecretive condition (as defined by need for two or more broncoaspirations per hour in the previous 8 hours) will be considered eligible. Patients will be excluded if contro-indications to High Frequency Percussive Ventilation and/or Electrical Impedance Tomography exist.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung aeration | Soon after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify the lung aeration (as assessed by the end-expiratory lung impedance through EIT), as compared to baseline before the treatment
Lung aeration | One hour after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify the lung aeration (as assessed by the end-expiratory lung impedance through EIT), as compared to baseline before the treatment
Lung aeration | Three hours after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify the lung aeration (as assessed by the end-expiratory lung impedance through EIT), as compared to baseline before the treatment

SECONDARY OUTCOMES:
Arterial Blood Gases | Soon after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify Arterial Blood Gases, as compared to baseline before the treatment
Arterial Blood Gases | One hour after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify Arterial Blood Gases, as compared to baseline before the treatment
Arterial Blood Gases | Three hours after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify Arterial Blood Gases, as compared to baseline before the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be shared after study publication on a peer-reviewed journal in english language, on a reasonable request to the principal investigator
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After study publication on a peer-reviewed journal in english language
Access Criteria: On reasonable request to the Principal Investigator

REFERENCES:
- [Derived] Garofalo E, Rovida S, Cammarota G, Biamonte E, Troisi L, Cosenza L, Pelaia C, Navalesi P, Longhini F, Bruni A. Benefits of secretion clearance with high frequency percussive ventilation in tracheostomized critically ill patients: a pilot study. J Clin Monit Comput. 2023 Jun;37(3):911-918. doi: 10.1007/s10877-022-00970-7. Epub 2023 Jan 6. PMID 36607533